CLINICAL TRIAL: NCT02313311
Title: Study Embryos of IVF by Time-lapse System
Brief Title: Select Embryos by Time-lapse System for Single Embryo Transfer
Acronym: SETLSSET
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Li-jun Ding (Other)
Responsible Party: Sponsor-Investigator, Li-jun Ding, Gulou Hospital, Nanjing University
Organization: Nanjing University (Other)
Other Study IDs: LJ201102-BK20141087-BL2014003; LJ201102 (Other Grant/Funding Number: Jiangsu Province, China)
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Embryo
Keywords: Cleavage pattern, timing parameter, time-lapse
MeSH Terms: interventions — Time-Lapse Imaging

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: time-lapse imaging — Embryos are observed using time-lapse imaging (Primo Vision®). It is an incubator with a compact, sealed, and digitally inverted camera unit which can automatically acquire images.The system can record the actual developmental stage of the embryos, all the recorded images can be saved to be analyzed later using a special software program.

SUMMARY:
The objective of this study is to establish a hierarchical embryo selection process by using the time-lapse imaging (TLI), combining the embryo cleavage patterns and timing parameters.

DETAILED DESCRIPTION:
The embryos of patients undergoing in vitro fertilization (IVF) treatment is cultured to blastocyst stage and observed by TLI. The association of embryo cleavage patterns/timing parameters and good-quality blastocyst rates are evaluated by logistic regression and to establish a hierarchical embryo selection. The value of the selection process is assess by single embryo transfer (SET) on Day 3.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing assistant reproduction treatment

Exclusion Criteria:

* Oocyte donation cycles

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing assistant reproduction treatment
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
good-quality blastocyst rate | 6 days post insemination

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, Dr., Principal Investigator — Reproductive Medicine Centre, Drum Affiliated to Hospital Nanjing University Medical School